CLINICAL TRIAL: NCT04276636
Title: Exploring the Effects of Caltrate Supplement on the Chronic Course of Crohn's Disease Patients With Vitamin D Deficiency，a Prospective Cohort Study
Brief Title: Exploring the Effects of Caltrate Supplement on the Chronic Course of Crohn's Disease Patients With Vitamin D Deficiency
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2020-01-102
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Crohn's Disease; Vitamin D Deficiency; Vitamin D Supplement
MeSH Terms: conditions — Crohn Disease; Vitamin D Deficiency | interventions — Calcium Carbonate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caltrate (Experimental): This group of patients are going to supplemented with Caltrate 0.6 g / d orally.
  Interventions: Drug: Caltrate Pill
- Control (No Intervention): The other group do not interfere.

INTERVENTIONS:
Drug: Caltrate Pill — Vitamin D-deficient CD patients are divided into two groups, one group is given orally with Caltrate Pill 0.6 g / d, while the other group do not interfere.
  Arms: Caltrate

SUMMARY:
Aims:Prospectively observe the effects of Caltrate supplementation on the chronic course of Crohn's disease patients, analyze whether the effect of Caltrate on CD patients is affected by factors such as disease site, disease activity, treatment, etc.Provide a certain theoretical basis for "precision treatment" for CD patients in the future.

Design：It is a prospective cohort study. Investigators include a total of 60 participants with CD according to the inclusion and exclusion criteria, and divide them into two groups to assess their initial disease activity and detect related indicators. At the same time，Investigators detect the Vitamin D Gene gene polymorphisms in all participants.One group is given Caltrate 0.6g per day orally, and the control group do not intervene. After 12 months, re-evaluate the disease activity and retest the relevant indicators, and use statistical methods to analyze whether Caltrate supplementation treatment can increase the serum 25 (OH) D level of CD participants, improve the condition of CD participants,relationship with Vitamin D Gene Polymorphism，and analyze the effect of Caltrate on participants with CD is affected by factors such as disease site, disease activity, and treatment.

DETAILED DESCRIPTION:
1. The research can be started only after approval by the Medical Ethics Committee of the Second Affiliated Hospital of Wenzhou Medical University.
2. According to the "Consensus on Diagnosis and Treatment of Inflammatory Bowel Disease" formulated by the Beijing Conference in 2018 as a standard, patients with clear diagnosis of CD are collected. Exclusion criteria included pregnancy, breastfeeding, liver and kidney dysfunction, concurrent autoimmune diseases, and use of antiepileptic drugs or drugs metabolized by liver cytochrome P450 enzymes.
3. Assess disease activity of CD participants based on the "Simplified Crohn's disease Activity Score".
4. General information about participants with CD is collected.
5. Detection of VDR gene polymorphisms using Snapshot technology.
6. Serum C-reactive protein, erythrocyte sedimentation rate, white blood cells, albumin, creatinine, alanine aminotransferase, calcium and phosphorus levels are measured.
7. The level of serum 25 (OH) D of participants is detected.
8. Develop a treatment plan for participants.
9. Participants are divided into two groups, one group is given oral Caltrate 0.6g / d, and the other group did not intervene.
10. The above serum indicators are re-measured in the 12th month, and the condition of CD participants is also evaluated.
11. Follow-up for 12 months. By comparing the above indicators, observe that in the Han population:

    1. Can Caltrate supplementation increase serum 25 (OH) D levels in patients with CD?
    2. Can Caltrate supplementation improve the condition of patients with CD?
    3. whether vitamin D gene polymorphisms affect the efficacy of Caltrate supplementation therapy?
    4. Analyze whether the effect of Caltrate on CD patients is affected by factors such as disease site, disease activity, treatment, etc ..
12. Through statistical analysis, comprehensive analysis of the effectiveness and safety of Caltrate supplementation in Han patients with CD, and its relationship with vitamin D gene polymorphisms, providing a theoretical basis for further "precise treatment" intervention in inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Clearly diagnosed patients with CD
* Vitamin D deficiency (<= 20ng / ml)

Exclusion Criteria:

* Pregnancy, lactation
* Liver and kidney insufficiency
* Co-morbid with other autoimmune diseases
* Use antiepileptic drugs or drugs metabolized by liver cytochrome P450 enzymes
* Vitamin D level is normal or high

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Serum 25 (OH) D level | 1year
  Because serum 25 (OH) D levels are relatively stable, they are considered the most reliable indicator of vitamin D status.

SECONDARY OUTCOMES:
White blood cell count | 1year
  White blood cell count can be used to reflect the degree of inflammation in the body
erythrocyte sedimentation rate | 1year
  ESR can be used to reflect the degree of inflammation in the body.
C-reactive protein. | 1year
  C-reactive protein can be used to reflect the degree of inflammation in the human body

CONTACTS AND LOCATIONS:
Overall Officials: Xia Xia long, Master, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- SAHWenzhouMU, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Data sets will be made available on relevant requests and in accordance with journal guidelines when publishing results from this study.